CLINICAL TRIAL: NCT04700683
Title: Chronic Efficacy and Usability of Transcutaneous Electrical Nerve Stimulation in Subjects With Restless Leg Syndrome (RLS)
Brief Title: Noninvasive Peripheral Nerve Stimulation for Restless Legs Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RLS-SNS01
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Noninvasive Peripheral Nerve Stimulation (Active Comparator): NPNS device programmed to deliver active stimulation.
  Interventions: Device: Noctrix Health NPNS device v1.0 - Active
- Sham control (Sham Comparator): NPNS device programmed to deliver sham stimulation.
  Interventions: Device: Noctrix Health NPNS device v1.0 - Sham

INTERVENTIONS:
Device: Noctrix Health NPNS device v1.0 - Active — Wearable device programmed to deliver electrical stimulation to peripheral nerves of the lower limbs.
  Arms: Noninvasive Peripheral Nerve Stimulation
Device: Noctrix Health NPNS device v1.0 - Sham — Wearable device programmed to deliver sham stimulation.
  Arms: Sham control

SUMMARY:
Prospective multi-site randomized sham-controlled crossover feasibility study evaluating tolerability and efficacy of noninvasive peripheral nerve stimulation (NPNS) for patients with moderate-severe primary Restless Legs Syndrome (RLS). Response to NPNS investigational device was compared to sham control in a 2x2 crossover design such that subjects were assigned to receive 2 weeks of NPNS and 2 weeks of sham, in randomized order.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate-severe RLS symptoms as defined by a score of 15 or greater points on IRLS.
* RLS symptoms are primarily noticeable in the subject's lower legs and/or feet.
* Subject reports having a medical diagnosis of primary idiopathic restless legs syndrome (RLS) or Willis-Ekbom Disorder (WED) OR Investigator has diagnosed the subject with primary idiopathic restless legs syndrome (RLS) or Willis-Ekbom Disorder (WED).
* Subject has experienced RLS symptoms at night on 2 or more nights per week during the previous month.
* On typical dose and schedule of RLS medication (if any), subject typically experiences RLS symptoms on 2 or more nights per week.
* RLS symptoms are primarily in the evening and night.
* Subject owns the necessary equipment to respond to texts, phone calls, and video calls.
* Subject is 18 years of age or older when written informed consent is obtained.
* Subject has signed a valid, Institutional Review Board (IRB)-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English.

Exclusion Criteria:

* Subject has RLS that is known to be caused by another diagnosed condition.
* Subject has active implantable medical devices anywhere in the body (including pacemakers), or passive medical devices implanted in the leg.
* Subject has an uncontrolled sleep disorder other than RLS that significantly interferes with their sleep as determined by the trial director or physician.
* Subject has been diagnosed with one of the following conditions: Epilepsy or other seizure disorder, Cellulitis or open sores of the legs, Renal failure, Iron-Deficiency Anemia, Severe movement disorder symptoms (Parkinson's disease, Huntington's disease, dyskinesia, dystonia), Deep Vein Thrombosis, Stage 4-5 Chronic Kidney Disease, Multiple sclerosis, Current, active or acute or chronic infection other than viral upper respiratory tract infections, A malignancy within the past 5 years (not including basal or squamous cell skin cancer)
* Subject is on dialysis or anticipated to start dialysis while participating in the study
* Subject is allergic to electrode gel, polyurethane foam, or lycra.
* Subject has severe edema in lower legs.
* Subject has failed a nerve conduction study prescribed by a physician or has been diagnosed with severe peripheral neuropathy.
* During Visit 1, subject cannot notice the stimulation at the maximal dose or cannot tolerate the stimulation at the minimal effective dose
* Subject selects Statement 2 or is unable to decide which of the following two statements most closely describe their condition: Statement 1: My symptoms are best characterized by a strong or overwhelming urge to move my legs. Moving my legs often results in temporary relief of that urge. Statement 2: My symptoms are best characterized by involuntary leg spasms that happen at regular intervals. These leg spasms can wake me up in the middle of the night."
* Subject has significantly changed medication dose or schedule of antidepressants, sleep medications, or RLS medications within the past 30 days.
* Recent history of alcohol or recreational drug abuse (within the past 6 months).
* Subject has received an investigational drug or device within the last 30 days or is planning to receive an investigational device during the duration of the study.
* Subject has undergone a major surgery (excluding dental work) in the previous 30 days.
* Subject has another medical condition that may affect validity of the study or put the subject at risk as determined by the investigator.
* Subject is unable or unwilling to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the clinical tolerability, usability, and patient response for the prototype device, with the intention of improving overall device performance. | Weeks 1-2 of each intervention
  Subject satisfaction and usability questionnaire

SECONDARY OUTCOMES:
Change from baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) score at week 2 | Week 2 of each intervention compared to week prior to study entry
  International Restless Legs Syndrome Study Group Rating Scale is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe.
Change to Summary NRS score of RLS symptom severity | Weeks 1-2 of each intervention
  Participant rating of average RLS symptom severity from 0-10 on a Numerical Rating Scale (NRS) scale, where 10 is the most severe. Participants complete a single Summary NRS scale at the end of each 2-week intervention, rating the average RLS symptoms before, during, and after device usage.
Change to Daily NRS score of RLS symptom severity | Weeks 1-2 of each intervention
  Participant rating of average RLS symptom severity from 0-10 on a Numerical Rating Scale (NRS) scale, where 10 is the most severe. Participants complete the Daily NRS scale each day during each 2-week intervention, rating the RLS symptoms before, during, and after the previous night of device use.
Responder rate on CGI-I scale at week 2 relative to baseline | Week 2 of each intervention compared to week prior to study entry
  Responder rate is defined as the proportion of responses of "Much Improved" or "Very Much Improved" relative to baseline on the 7-point participated-rated Clinical Global Impressions-Improvement (CGI-I) scale.

OTHER OUTCOMES:
Change to NRS score of RLS severity during SIT procedure | During the 60 minute SIT procedure
  The 60-minute Suggested Immobilization Test (SIT) assesses RLS symptom severity in a controlled procedure in the following three conditions: no device, NPNS device, Sham device. At SIT start and after every 10 minutes, the participant rates average RLS symptom severity from 0-10 on a Numerical Rating Scale (NRS) scale, where 10 is the most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Charlesworth, PhD, Study Director — Noctrix Health, Inc.
Locations (3):
- United States (3):
  - Mark J Buchfuhrer private practice, Downey, California
  - SRI International Human Sleep Research Lab, Menlo Park, California
  - Sleep Medicine Specialists of California, San Ramon, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charlesworth JD, Adlou B, Singh H, Buchfuhrer MJ. Bilateral high-frequency noninvasive peroneal nerve stimulation evokes tonic leg muscle activation for sleep-compatible reduction of restless legs syndrome symptoms. J Clin Sleep Med. 2023 Jul 1;19(7):1199-1209. doi: 10.5664/jcsm.10536. PMID 36856064
- [Derived] Buchfuhrer MJ, Baker FC, Singh H, Kolotovska V, Adlou B, Anand H, de Zambotti M, Ismail M, Raghunathan S, Charlesworth JD. Noninvasive neuromodulation reduces symptoms of restless legs syndrome. J Clin Sleep Med. 2021 Aug 1;17(8):1685-1694. doi: 10.5664/jcsm.9404. PMID 33949942